CLINICAL TRIAL: NCT00935571
Title: Incidence of Postthoracotomy Pain Following General Anesthesia: A Comparison Between TIVA and Inhalation Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: In Cheol Choi, Asan Medical Center
Other Study IDs: 20090708
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Lung Cancer; Neoplasms, Lung
MeSH Terms: conditions — Lung Neoplasms | interventions — Propofol; Remifentanil; Sevoflurane

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group I, Group II: Group I: anesthetized with TIVA (Propofol + Remifentanil)
  Group II: anesthetized with inhalation (sevoflurane)
  Interventions: Drug: propofol, remifentanil, sevoflurane

INTERVENTIONS:
Drug: propofol, remifentanil, sevoflurane — Propofol: using target controlled infusion (TCI); 1-3ug/ml remifentanil: using TCI by 5-20 ng/ml sevoflurane: 2-3volume% (1-2 MAC)
  Other Names: diprivan; ultiva

SUMMARY:
The purpose of this study is to evaluate the incidence of postthoracotomy pain between total intravenous anesthesia (TIVA)and inhalation anesthesia after lung surgery.

DETAILED DESCRIPTION:
Thoracotomy is one of the most painful surgical incisions. It has been shown that 5-80% of patients still suffer from thoracic pain 2-3 months after surgery and the international association for the study of pain (IASP) defines postthoracotomy pain syndrome (PTTS)as pain that recurs or persists at least 2 months after surgical procedure. Previous reports have shown that the incidence of PTTS varies according to preoperative pain, pain intensity, sex, and types of procedure. However, little is known about the effect of the type of anesthesia to postthoracotomy pain.

ELIGIBILITY:
Inclusion Criteria:

* patients undergo elective thoracotomy of lung surgery

Exclusion Criteria:

* emergency operation age under 18 years patients with unstable hemodynamics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled to undergo elective thoracotomy of lung surgery
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-06 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of pain | 3 and 6 months later after operation

SECONDARY OUTCOMES:
pain characters | 3 and 6 months later after operation

CONTACTS AND LOCATIONS:
Overall Officials: In Cheol Choi, MD, PhD, Study Chair — Department of Anesthesiology and Pain Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Gotoda Y, Kambara N, Sakai T, Kishi Y, Kodama K, Koyama T. The morbidity, time course and predictive factors for persistent post-thoracotomy pain. Eur J Pain. 2001;5(1):89-96. doi: 10.1053/eujp.2001.0225. PMID 11394926